CLINICAL TRIAL: NCT03586856
Title: Trial of NCPAP Interface Leakage (ToNIL): A Randomised Crossover Comparison of Leakage With Nasal Prongs and Nasal Mask Interface in Newborn Infants Treated With CPAP
Brief Title: Comparison of Leakage With Nasal Prongs and Nasal Mask Interface in Newborns Receiving CPAP Treatment
Acronym: ToNIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baldvin Jonsson (Other)
Responsible Party: Sponsor-Investigator, Baldvin Jonsson, Associate Professor, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2016/2449-31
Record Dates: First submitted 2018-06-04; First posted 2018-07-16 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Respiration; Insufficient or Poor, Newborn; Infant,Premature
Keywords: Continuous positive airway pressure; Air Leakage; Work of breathing
MeSH Terms: conditions — Respiratory Aspiration; Premature Birth

STUDY DESIGN:
Intervention Model Description: Main study design: Two armed randomized cross-over comparison of leakage for two interfaces. The trial also investigates simple measures to reduce leakage (observational)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nasal mask interface (Active Comparator): The CPAP interface will be applied and adjusted by experienced staff blinded to the outcome variable; leakage. Measures to reduce/minimize leakage are tested in an unblinded observational part after the intervention.
  Interventions: Device: Nasal mask interface
- Nasal prongs interface (Active Comparator): The CPAP interface will be applied and adjusted by experienced staff blinded to the outcome variable; leakage. Measures to reduce/minimize leakage are tested in an unblinded observational part after the intervention.
  Interventions: Device: Nasal prongs interface

INTERVENTIONS:
Device: Nasal mask interface — Nasal masks is a standard interface used for CPAP treatment of newborn infants. The CPAP device allows for easily switching between the nasal prongs or nasal mask interface as well as adjustment of size.
  Arms: Nasal mask interface
Device: Nasal prongs interface — Nasal masks is a standard interface used for CPAP treatment of newborn infants. The CPAP device allows for easily switching between the nasal prongs or nasal mask interface as well as adjustment of size.
  Arms: Nasal prongs interface

SUMMARY:
The study is a two-armed randomized cross-over comparison of leakage with nasal prongs and nasal mask interface in newborn infants treated with CPAP, born after 28 weeks of gestational age. For infants with an interface leakage, the trial also includes an observational part evaluating simple measures to reduce leakage.

The study will be carried out in the Karolinska University Hospital Stockholm and in the Östersund Hospital.

DETAILED DESCRIPTION:
The study will recruit a total of 50 infants receiving CPAP for respiratory support at the Karolinska University Hospital and the Östersund Hospital. The infant should be stable and not in major respiratory distress. Consent from the parents will be obtained before enrolment.

The included infants should have stable spontaneous breathing and be older than 28 weeks (corrected age) at the time of enrolment. The reason for respiratory failure and CPAP treatment is not relevant for study purposes. If an infant cannot participate in the study at a given time, he or she can be enrolled later. A child can only participate once.

The primary outcome is leakage. This is recorded using equipment for measuring air flow during CPAP treatment. Measurement of leakage is first performed for one interface and then the next (cross-over). The interface order is randomized. The leakage will be measured after a few minutes of stabilization (part 1). If there is leakage, a few simple measures to reduce the leakage will be evaluated (part 2). The second part will approximately add 10-20 minutes and includes simple measures such as adjusting the nasal mask, closing the mouth, changing the position or changing the size of nasal mask/prongs. Part 1 and part 2 are then repeated for the next interface. If the child shows signs of distress or agitation the measurement will be paused or stopped.

Part 1: The CPAP system with the randomized interface (nasal mask or nasal prongs) is applied and adjusted by experienced NICU staff. The staff is blinded for the outcome variable, leakage. The choice of size and other adjustments are guided by clinical experience and not by protocol. The NICU staff is not allowed to participate in the explorative part where measures to reduce leakage are evaluated. This precaution is to avoid staff learning what adjustments affect leakage and influence care of infants enrolled at a later stage.

Part 2: In this part the investigators can evaluate the effect of simple measures to minimize the leakage. The level of leakage is displayed on a screen. Examples of measures are; closing the mouth of the infant, adjusting straps, adjusting position and changing the size of the interface. Not every child will undergo all measures to reduce leakage, since the aim of this explorative part is to explore ways to reduce leakage.

It is estimated that these tests and measures will take 15-60 minutes per child. No other measurements or follow-up is planned. No blood samples will be collected or analysed.

The study will collect information on the infant and the birth. This includes birth weight, gestational age at birth, gender, previous respiratory support and medical history.

The main outcome variable is absolute leakage (via mouth or via CPAP interface). Other collected variables are oxygen saturation, respiratory rate, inspired oxygen concentration, apneas, heart rate, if the infant is awake/asleep or in distress. Safety variables include skin irritation or damage of the nose caused by the interface, instability or deterioration of respiration or circulation, problems with the equipment or other adverse events. The investigation can be stopped immediately in the case of distress or instability. The study is, as far as the investigators know, the first one of its kind. The air flow meters do not affect the CPAP system and use a technique that measures the total leakage in L/min. These improvements have been emphasized in previous studies. The study follows GCP (good clinical practice) standards and The Helsinki declaration.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age over 28 weeks (corrected age) at the time of inclusion
* Patient receiving respiratory support with CPAP

Exclusion Criteria:

* Airway, pulmonary, cardiac or gastro-intestinal malformations
* Neuromuscular disease
* Circulatory unstable patient
* FiO2 higher than 0.5
* Nasal damage or major skin irritation.
* Extubation less than 24 h before investigation
* Surgery less than 5 days before investigation

Max Age: 44 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-10-26 (Actual); Study Completion 2019-10-26 (Actual)

PRIMARY OUTCOMES:
Leakage in the CPAP system | 0-60 min
  Measurement of absolute leakage (at interface or mouth) using flowmeters connected to the CPAP device in flow through position (L/min, 30 seconds recording)

SECONDARY OUTCOMES:
Inspired oxygen level (FiO2) | 0-60 min
  FiO2 level and adjustments needed to maintain pre-intervention baseline peripheral oxygen saturation (SpO2 target range according to local guidelines)
Level of CPAP support (cmH2O) | 0-60 min
  CPAP level and adjustments needed to maintain pre-intervention baseline peripheral oxygen saturation (SpO2 target range according to local guidelines)
Peripheral oxygen saturation (SpO2) | 0-60 min
  Deviations from baseline and changes requiring adjustment of respiratory support (Outcome 2 and 3)
Measurement completion possible (yes/no) | 0-60 min
  The number of infants (ratio of total included patients) where measurement of leakage could be determined (on first or more attempts)
Effect of simple measures to reduce leakage (L/min) | 0-60 min
  Lowest level of recorded level of leakage obtainable using simple measures to reduce leakage, guided by leakage monitoring equipment (L/min and measures used to achieve reduction)

OTHER OUTCOMES:
Safety variable: Desaturation during measurement | 0 to competition of measurement (maximum 3 hours)
  Desaturation (SpO2) from baseline requiring treatment or adjustment, during manipulation or leakage measurement.
Safety variable: Apneas during measurement | 0 to competition of measurement (maximum 3 hours)
  Apneas requiring treatment or adjustment, during manipulation or leakage measurement.
Safety variable: FiO2 adjustments during measurement | 0 to competition of measurement (maximum 3 hours)
  FiO2 adjustments required, during manipulation or leakage measurement.
Safety variable: Circulatory instability | 0 to competition of measurement (maximum 3 hours)
  Circulatory instability (bradycardia or hypotension) requiring treatment or adjustment, during manipulation or leakage measurement.
Safety variable: Nasal irritation | 0 to competition of measurement (maximum 3 hours)
  Nasal irritation requiring treatment or attention, during or after manipulation and leakage measurement.
Safety variable: Pneumothorax | 0 to competition of measurement (maximum 3 hours)
  Confirmed pneumothorax or air-leak, during manipulation or leakage measurement.
Safety variable: Adverse events | 0 to competition of measurement (maximum 3 hours)
  Problems related to trial or equipment used, classified as adverse events according to GCP (Good Clinical Practice)
Safety variable: Adherence to protocol | 0 to competition of measurement (maximum 3 hours)
  Problems related to following study protocol
Safety variable: Problems with equipment | 0 to competition of measurement (maximum 3 hours)
  Problems related to study equipment

CONTACTS AND LOCATIONS:
Overall Officials: Baldvin Jonsson, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Östersund hospital, Östersund, Jämtland County
  - Karolinska University Hospital, Neonatology department, Stockholm

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gunnarsdottir K, Falk M, Baldursdottir S, Donaldsson S, Jonsson B, Drevhammar T. Do newborn infants exhale through the CPAP system? Secondary analysis of a randomised cross-over trial. Arch Dis Child Fetal Neonatal Ed. 2023 May;108(3):232-236. doi: 10.1136/archdischild-2022-324462. Epub 2022 Oct 19. PMID 36261145